CLINICAL TRIAL: NCT07108712
Title: The Role of Diffusion Magnetic Resonance Imaging (dMRI) in the Early Evaluation of Brain White Matter Diseases
Brief Title: Diffusion Magnetic Resonance Imaging (dMRI) in the Early Evaluation of Brain White Matter Diseases
Status: Recruiting | Type: Observational
Sponsor: The General Authority for Teaching Hospitals and Institutes (Network)
Responsible Party: Principal Investigator, Hekmat Samir Baumey, Lecturer of Diagnostic Radiology, Damnhour National Medical Institute, The General Authority for Teaching Hospitals and Institutes
Other Study IDs: HD000235
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Diffusion Magnetic Resonance Imaging; Brain White Matter Diseases
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients diagnosed with suspected early-stage white matter disease (e.g., multiple sclerosis, small vessel disease, Alzheimer's disease, frontotemporal dementia, leukoaraiosis) will be enrolled.
  Interventions: Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Imaging (MRI) Scanner: All imaging will be performed using a 1.5 tesla MRI scanner to ensure high resolution and signal-to-noise ratio.

SUMMARY:
To assess the sensitivity and accuracy of diffusion magnetic resonance imaging (MRI), including diffusion-weighted imaging (DWI) metrics, in identifying early-stage changes in brain white matter related to various white matter diseases.

DETAILED DESCRIPTION:
Brain white matter diseases (WMDs) are a group of neurological conditions that involve changes to the brain's white matter, often leading to cognitive, motor, and sensory impairments.

Diffusion Magnetic Resonance Imaging (dMRI), has emerged as a powerful non-invasive imaging tool for evaluating microstructural changes in brain white matter. This protocol aims to investigate the role of dMRI in the early identification and characterization of brain white matter diseases, focusing on its potential for detecting abnormalities before the onset of overt clinical symptoms.

Diffusion-weighted imaging (DWI), one of the first advanced magnetic resonance imaging (MRI) techniques, has rapidly ascended on the basis of its applicability in strokes and some infectious diseases. Restricted diffusion is significant information in the context of vascular ischemia, helping to delimit the brain-damaged area

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years.
* Clinical suspicion of early-stage white matter disease.
* No prior diagnosis of significant neurological disorders (e.g., stroke, brain tumors).
* Ability to provide informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Contraindications for magnetic resonance imaging (MRI) (e.g., metal implants, pacemakers).
* Severe psychiatric or cognitive impairment that prevents participation.
* Control Group: Healthy individuals without any clinical history of neurological diseases, matched by age and sex to the patient cohort.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be a multicenter, cross-sectional study will be conducted on patients diagnosed with suspected early-stage white matter disease (e.g., multiple sclerosis, small vessel disease, Alzheimer's disease, frontotemporal dementia, leukoaraiosis) will be enrolled. Healthy age-matched controls will also be included for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of diffusion magnetic resonance imaging | Immediately after diffusion magnetic resonance imaging (Up to 1 hour)
  Sensitivity of diffusion magnetic resonance imaging to predict the early evaluation of brain white matter diseases

CONTACTS AND LOCATIONS:
Locations (1):
- General Authority for Teaching Hospitals and Institutes, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.